CLINICAL TRIAL: NCT00865176
Title: Comparative Bioavailability Study of Eplerenone 50 mg Tablets (Sandoz Inc., USA) and Inspra 50 mg Tablets (GD Searle LLC, USA) in Healthy Male and/or Female Volunteers Under Fasting Conditions.
Brief Title: Comparative Bioavailability Study of Eplerenone 50 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P1DX06002
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2009-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Eplerenone

ARMS (2):
- 1 (Experimental): Eplerenone 50mg Tablets
  Interventions: Drug: Eplerenone 50 mg Tablets Sandoz Inc., USA
- 2 (Active Comparator): INSPRA 50mg Tablets
  Interventions: Drug: Inspra 50 mg Tablets GD Searle LLC, USA

INTERVENTIONS:
Drug: Eplerenone 50 mg Tablets Sandoz Inc., USA
  Arms: 1
Drug: Inspra 50 mg Tablets GD Searle LLC, USA
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the relative bioequivalence of Eplerenone 50 mg ER Tablets under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2006-06; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Bioequivalence according to US FDA guidelines | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Deepen Patel, M.D., CCFP, Principal Investigator — Allied Research International Inc.